CLINICAL TRIAL: NCT03525535
Title: MeAsurement of uneXpected Acute Pulmonary embolIsM Among Not Anticoagulated Patients Older Than 75 Years Admitted With Syncope.
Brief Title: Prevalence Rate of Pulmonary Embolism Among Not Anticoagulated Patients
Acronym: MAXIME
Status: Terminated | Type: Observational
Why Stopped: Principal investigator departure without possible replacement
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-CHITS-04; 2017-A01197-46 (Other: Id-RCB)
Record Dates: First submitted 2018-05-03; First posted 2018-05-15 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary embolism: data from routine care will be collected for patient eligible and willing to participate
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — data from patient included will be collected during the study

SUMMARY:
The purpose of this study is to evaluate the prevalence rate of pulmonary embolism among not anticoagulated patient older than 75 years old admitted with syncope and hospitalised in the Toulon Hospital

DETAILED DESCRIPTION:
This study will be proposed to every patient that correspond to eligibility criteria. Will be included only those who are not opposed to the collection of their data.

The data collected will come from the routine care such as medical history, clinical datas, imaging data… The number of pulmonary imaging will be assessed before the diagnostic strategy proposed by Dr Prandoni and after the application of this strategy thanks to a questionnaire to physicians.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female over 75 years-old
* Emergency consult resulting on an hospitalization in the geriatric service or in the internal medicine service
* Hospitalised in the Centre Hospitalier Intercommunal de Toulon for syncope, presenting these symptoms:
* Loss of consciousness with quick return to normal (less than one minute)
* Spontaneous resolution

Exclusion Criteria:

* history of syncope
* other loss of consciousness (epilepsy, stroke, head trauma)
* anticoagulated treatment
* patient's objection

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: male or female over 75 years old without anticoagulated treatment hospitalized for syncope symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Pulmonary embolism prevalence | 24 month
  Prevalence rate of pulmonary embolism among patient hospitalized for syncope and diagnosed with ventilation/perfusion scan or CT scan.

SECONDARY OUTCOMES:
Assess the impact of the Prandoni's recommendations on the paraclinical evaluations | 24 month
  Number of CT-scans that are made systematically since the Prandoni's recommendations are applied in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Faucher, MD, Principal Investigator — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (1):
- Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, La Seyne-sur-Mer, Var, France

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD